CLINICAL TRIAL: NCT01219192
Title: Phase I Study of M2ES in Patients With Advanced Pancreatic Cancer After Gemcitabine Treatment Failure
Brief Title: Study of M2ES in Patients With Advanced Pancreatic Cancer After Gemcitabine Treatment Failure
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Protgen Ltd (Industry)
Responsible Party: Guodong CHANG, Protgen Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2ES2010-2
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2010-10-28 (Estimated); Status verified 2010-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- M2ES 15mg (Experimental)
  Interventions: Drug: M2ES
- M2ES 30mg (Experimental)
  Interventions: Drug: M2ES
- M2ES 45mg (Experimental)
  Interventions: Drug: M2ES
- M2ES 60mg (Experimental)
  Interventions: Drug: M2ES 60mg

INTERVENTIONS:
Drug: M2ES — M2ES IV D1,8,15,21 every 28 days a cycle
  Other Names: M2ES 15mg intervention
  Arms: M2ES 15mg
Drug: M2ES — M2ES IV D1,8,15,21, every 28days a cyce.
  Other Names: M2ES 30mg intervention
  Arms: M2ES 30mg
Drug: M2ES — M2ES 45mg IV D1,8,15,22 28days a cycle
  Other Names: M2ES 45mg intervention
  Arms: M2ES 45mg
Drug: M2ES 60mg — M2ES 60mg IV D1,8,15,22 every 28days a cycle
  Other Names: M2ES 60mg intervention
  Arms: M2ES 60mg

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability and determine the recommended dosing for the treatment in patients with advanced pancreatic cancer after fist-line Gemcitabine treatment failure.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability and determine the recommended dosing for the treatment in patients with advanced pancreatic cancer after fist-line Gemcitabine treatment failure.We star with the dose M2ES 15mg,then escalate to 30mg 45mg 60mg,to find the recommended dose in clinic practise.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically confirmed pancreatic adenocarcinoma that was not amenable to potentially curative surgery.
2. All patients must have developed progressive disease (PD) while receiving or within 6 months after discontinuing palliative gemcitabine-based chemotherapy
3. Prior radiation therapy was allowed provided that the only sites of measurable disease were not located within the radiation port.
4. 18 years of age or older
5. Karnofsky performance status (KPS) of 60-100 points
6. measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
7. Adequate hematologic, renal, and hepatic function was required as deWned by the following: WBC ≥3.5×109/L, absolute neutrophil count ≥ 1.5 × 109/L, platelet count ≥100 × 109/L, hemoglobin≥9g/dL, total bilirubin ≤2.5 upper limit of normal [ULN],AST≤2.5 ULN, or≤5 ULN if there was evidence of liver metastases;alkaline phosphatase≤ 2.5 ULN, or≤ 5 ULN if there was evidence of liver Metastases creatinine clearance≤50 mL/min,
8. life expectancy of at least 12 weeks

Exclusion Criteria:

1. patients had clinically apparent CNS metastases or carcinomatous meningitis
2. another active malignancy, or any history of other malignancy within the past 5 years except for nonmelanoma skin cancer and carcinoma in situ of the cervix
3. more than 3 weeks intervals between the last administration of the prior chemotherapy regimen and study entry
4. more than 4 weeks intervals between the last administration of the targeted therapy regimen and study entry
5. major surgery within the prior 6 weeks;
6. Pregnant or lactating women
7. tumor involvement of major blood vessels
8. uncontrolled intercurrent illness
9. A history of myocardial infarction or stroke within the last 6 months, uncontrolled hypertension, unstable angina
10. clinically significant cardiac disease (eg, congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication, or myocardial infarction)
11. urine protein ≥ 500 mg in 24 hours;
12. evidence of bleeding diathesis or coagulopathy
13. Patients on therapeutic doses of low-molecular weight heparin
14. Patients who received thrombolytic agents within the previous month or who required full-dose anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
MDT | 3 weeks
  The maximum tolerable dosage

SECONDARY OUTCOMES:
PFS | 4 months
  progress free survival

CONTACTS AND LOCATIONS:
Overall Officials: Shunchang JIAO, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China